CLINICAL TRIAL: NCT00092937
Title: Secondary Transplantation Using Moderate Dose Busulfan as Conditioning for a Patient With Partial Reconstitution Post Initial Allogeneic Transplantation
Brief Title: Use of Busulfan as Conditioning Agent for a Second Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Elizabeth M. Kang, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040289; 04-I-0289
Record Dates: First submitted 2004-09-24; First posted 2004-09-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-04-06

CONDITIONS: Granulomatous Disease; Chronic
Keywords: Chronic Granulomatous Disease; Nonmyeloablative; CD34 Positive Cells; Donor Engraftment; Myeloid Chimerism
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Granulomatous Disease, Chronic | interventions — Busulfan

INTERVENTIONS:
Drug: Busulfan

SUMMARY:
This protocol is designed for a single specific patient. It uses busulfan as a conditioning agent in a second stem cell transplant procedure for a patient with chronic granulomatous disease (CGD), a disorder in which a certain type of white cells, called myeloid cells, do not function properly. This causes increased risk of serious bacterial and fungal infections that can lead to organ dysfunction, such as kidney disease, as well as formation of granulomas-non-cancerous masses that can cause obstructions in the esophagus, stomach, and intestines, and block urine flow from the kidneys and bladder.). The child in this study has previously undergone a stem cell transplant to treat CGD, and, as a result, he is now producing normal lymphocytes (another type of white cell). However, the myeloid cells from the donor did not engraft successfully, and the patient is still producing his own defective myeloid cells. In this study, the child will undergo a second stem cell transplant in combination with busulfan, a drug that targets myeloid cells, killing them to make way for healthy, donated myeloid cells.

Treatment includes the following procedures:

* Medical evaluation to confirm that the patient is healthy enough to undergo the transplantation
* Treatment with busulfan, injected through the patient's central venous line
* Stem cell transplantation through the central venous line
* Blood tests on days 25, 56, and 91 after the transplant to assess how many cells are of donor origin
* Bone marrow aspiration on day 100, and then at 12, 24, and 36 months to assess how many cells are of donor origin
* Pulmonary function (breathing) test at 12 and 24 months
* Physical examination and blood tests, weekly or twice weekly for the first 2 to 3 months and at 4, 6, 12, 18, 24, 36, 48, and 60 months after transplant
* Treatment for graft-versus-host disease (GVHD), if this complication develops. GVHD is the attack of lymphocytes from the donor against the patient's own cells. This is good if it is against abnormal cells, but bad if serious damage occurs to the patient's vital organs. GVHD is treated with steroids and cyclosporine, and possibly other drugs if needed.

DETAILED DESCRIPTION:
This is a single patient study using intravenous busulfan as a conditioning agent for a second allogeneic stem cell transplant in order to increase myeloid engraftment in a previously transplanted recipient with chronic granulomatous disease (CGD).

CGD is an inherited disorder of neutrophil function leading to increased risk of infections from both common and rare microorganisms, including fungi. Although these infections can often be prevented or successfully treated, there are long-term sequelae including organ dysfunction as a result of both the infections and the treatment. For example, many of the anti-fungal agents cause renal impairment and can even lead to kidney failure requiring dialysis. In addition, the abnormal functioning of the neutrophils leads to the development of granulomas, which can cause obstruction of various organs, in particular within the gastrointestinal and urogenital systems with sometimes serious sequelae. As a result the life expectancy of patients with CGD is significantly limited with no patients documented reaching the age of 50 and a 2 percent mortality rate per year of life.

Currently, the only available cure of CGD is bone marrow transplantation; however given its own inherent associated morbidities and mortality, as well as the necessity for a matched (related) donor, this has not been offered to all patients. More recently attempts to reduce the toxicities of this potentially curative treatment have lead to the development of non-myeloablative regimens, which as a result, can lead to partial engraftment of the donor cells into the recipient, a situation referred to as mixed chimerism. In order to achieve an adequate number of normal neutrophils for clinical benefit, the level of donor chimerism needs to be at least 5 percent in the myeloid lineage. One of the patients treated on a previous protocol with a novel nonmyeloablative conditioning regimen, has had 100 percent engraftment of his lymphoid cells, but less than 1percent engraftment of his myeloid lineage. As a result, he continues to experience the problems associated with CGD, but has had no problems of graft versus host disease (GVHD). In order to improve his myeloid engraftment, while taking advantage of the presence of his 100 percent lymphoid chimerism, we propose to treat him with moderate dose busulfan and a purified stem cell product from the original donor as a second transplant. With this study, the goal will be to improve this patient's myeloid engraftment so as to ostensibly cure him of his CGD.

ELIGIBILITY:
* RECIPIENT INCLUSION/EXCLUSION CRITERIA:
* The recipient fulfills by study design the inclusion criteria
* The patient however, would be considered ineligible for the study only If his donor is unable to participate.

DONOR EXCLUSION CRITERIA:

* Pregnant or lactating.
* Donor unfit to receive G-CSF and undergo apheresis. (Uncontrolled hypertension, history of congestive heart failure or unstable angina, thrombocytopenia).
* HIV positive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-09-23; Primary Completion 2010-04-06 (Actual); Study Completion 2010-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Winkelstein JA, Marino MC, Johnston RB Jr, Boyle J, Curnutte J, Gallin JI, Malech HL, Holland SM, Ochs H, Quie P, Buckley RH, Foster CB, Chanock SJ, Dickler H. Chronic granulomatous disease. Report on a national registry of 368 patients. Medicine (Baltimore). 2000 May;79(3):155-69. doi: 10.1097/00005792-200005000-00003. PMID 10844935
- [Background] Johnston RB Jr. Clinical aspects of chronic granulomatous disease. Curr Opin Hematol. 2001 Jan;8(1):17-22. doi: 10.1097/00062752-200101000-00004. PMID 11138621
- [Background] Roesler J, Brenner S, Bukovsky AA, Whiting-Theobald N, Dull T, Kelly M, Civin CI, Malech HL. Third-generation, self-inactivating gp91(phox) lentivector corrects the oxidase defect in NOD/SCID mouse-repopulating peripheral blood-mobilized CD34+ cells from patients with X-linked chronic granulomatous disease. Blood. 2002 Dec 15;100(13):4381-90. doi: 10.1182/blood-2001-12-0165. Epub 2002 Aug 1. PMID 12393624